CLINICAL TRIAL: NCT00583024
Title: Phase II Study of Adenovirus/PSA Vaccine in Men With Hormone - Refractory Prostate Cancer
Acronym: APP22
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David M Lubaroff (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, David M Lubaroff, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201705744; PC061667/2; 200605710 (Other: Initial UI IRB ID #)
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Hormone Refractory Prostate Cancer
Keywords: prostate cancer; vaccine; immunotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adenovirus/PSA Vaccine (Experimental): Participants will receive three injections of 0.16 ml. (0.125 ml. vaccine + 0.035 ml. Gelfoam) of the Ad/PSA subcutaneously
  Interventions: Biological: ADENOVIRUS/PSA VACCINE

INTERVENTIONS:
Biological: ADENOVIRUS/PSA VACCINE — 1x10E8 pfu in Gelfoam subcutaneously on days 0, 30, 60

SUMMARY:
This investigational study involves treatment with an Ad/PSA vaccine for men with prostate cancer who present with evidence of hormone refractory metastatic disease.

DETAILED DESCRIPTION:
Subjects in this trial will be eligible if they have recent evidence of hormone refractory disease (D3) and either (a) have a positive bone scan or a positive CT scan (with obvious soft tissue metastasis or lymph nodes >1 cm), with a PSA doubling time of >/= 12 months, a total PSA of < 5 mg/ml, and are asymptomatic; or (b) have a negative bone scan with any PSA doubling time, are asymptomatic, and are not a candidate for chemotherapy.

This is a virus vaccine in which the gene for prostate specific antigen (PSA) has been placed into a common cold virus termed adenovirus (Ad) to produce this Ad/PSA product. The purpose of this study is to determine whether vaccination with the Ad/PSA vaccine will induce an anti-PSA immunity that will result in the destruction of the remaining prostate cancer cells.

Subjects will be vaccinated three times, each injection administered at 30-day intervals. Based upon our earlier clinical trial, the vaccine is considered safe and should not induce any major side effects. The investigators hope that vaccination with this PSA virus will cause the body to produce immunity to the PSA and that immunity will destroy any cell that produces PSA. Since the only cells left in the body that produce PSA will be the cancer cells, the investigators propose that the vaccination and ensuing anti-PSA immunity will kill the prostate cancer cells. Importantly, this treatment should not cause any major side effects as would treatment with anti-cancer drugs.

ELIGIBILITY:
Inclusion criteria:

* Men with prostate cancer who present with evidence of hormone refractory disease (D3).
* Men with a positive bone scan or a positive CT scan (with obvious soft tissue metastasis or lymph nodes >1 cm), a PSA doubling time of >/= 6 months, and a total PSA of <10 ng/ml, and asymptomatic OR men with a negative bone scan and a negative CT scan with any PSA doubling time and asymptomatic.
* Scans must be obtained within 6 weeks of initiation of treatment.
* Written informed consent.
* Age >/= 18 years.
* Required laboratory values (obtained within 2 weeks of initiation of treatment)
* Serum creatinine </= 2.0 mg/dL
* Adequate hematologic function: granulocytes >/= 1800 per mm3, platelets >/= 100,000 per mm3, WBC >/= 3700, and lymphocytes >590.
* Adequate hepatocellular function: AST <3x upper limit of normal and total bilirubin <1.5 mg/dl (unless bilirubin elevation is consistent with Gilbert's syndrome).
* Castrate levels of testosterone of </= 50 ng/ml.
* PSA can be used as an eligibility criterion must be drawn within 28 days prior to injection number 1 and will be drawn on Day 1 for use as a baseline value.

Exclusion criteria:

* Active or unresolved clinically significant infection.
* Parenteral antibiotics <7 days prior to initiation of treatment.
* Evidence of prior or current CNS metastases. Specific imaging is not necessary in the absence of signs or symptoms.
* Co-morbid medical conditions which would result in a life expectancy (participation) of less than 1 year.
* Patients with compromised immune systems; congenital, acquired, or drug-induced (immunosuppressive agents) will be excluded from the study. Use of prednisone at doses higher than 10 mg daily (or equipotent steroid doses) for more than 7 days within 3 months of initiation of treatment is not allowed.
* Pre-existing malignancies that required treatment within the past 5 years except for basal or squamous cell cancers of the skin.
* Prior participation in any vaccine studies for non-infectious diseases.
* Prior chemotherapy, defined as prior cytotoxic chemotherapy for prostate cancer (or any cancer unless more than 5 years have elapsed). Examples of cytotoxic chemotherapy are mitoxantrone/prednisone and taxanes. Drugs such as Casodex or ketoconazole treatment must have been completed at least 6 weeks prior to initiation of treatment.
* The inability to understand the language and the clinical protocol.
* Allergy or religious objection to pork products; Gelfoam is produced from pork.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Lubaroff, PhD, Principal Investigator — University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elzey BD, Siemens DR, Ratliff TL, Lubaroff DM. Immunization with type 5 adenovirus recombinant for a tumor antigen in combination with recombinant canarypox virus (ALVAC) cytokine gene delivery induces destruction of established prostate tumors. Int J Cancer. 2001 Dec 15;94(6):842-9. doi: 10.1002/ijc.1556. PMID 11745487
- [Background] Lubaroff DM, Konety B, Link BK, Ratliff TL, Madsen T, Shannon M, Ecklund D, Williams RD. Clinical protocol: phase I study of an adenovirus/prostate-specific antigen vaccine in men with metastatic prostate cancer. Hum Gene Ther. 2006 Feb;17(2):220-9. doi: 10.1089/hum.2006.17.220. No abstract available. PMID 16454655
- [Result] Cavacini LA, Duval M, Eder JP, Posner MR. Evidence of determinant spreading in the antibody responses to prostate cell surface antigens in patients immunized with prostate-specific antigen. Clin Cancer Res. 2002 Feb;8(2):368-73. PMID 11839651

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adenovirus/PSA Vaccine
Started | 32
Completed | 28
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Adenovirus/PSA Vaccine
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stable, Decreased, or Increased PSA Doubling Times (PSADT)
Description: To evaluate the increase, decrease, or stable response rates (PSA responses and changes in PSADT) of the Ad/PSA vaccine using a prime-boost immunization strategy. PSADT will be calculated based on the MSKCC online calculator.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Adenovirus/PSA Vaccine
Number analyzed (Participants) | 26
Participants
  Decreased PSADT | 7
  Stable PSADT | 2
  Increased PSADT or PSA decline | 17

2. Primary Outcome: Number of Participants Who Develop a Strong or Modest Anti-PSA Immune Response
Description: Strong or modest antibody responses to PSA measured by the binding to PSA-secreting cell lines
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Adenovirus/PSA Vaccine
Number analyzed (Participants) | 25
participants
  Strong response | 15
  Modest response | 3

3. Secondary Outcome: Number of Participants Alive and Deceased Following Treatment
Description: To evaluate survival in evaluable patients receiving the Ad/PSA vaccine, as measured by 2-year, 5-year, 10-year, and overall survival (OS)
Time Frame: Every 6 months, up to 14 years
Population: 4 patients lost to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Adenovirus/PSA Vaccine
Number analyzed (Participants) | 28
Participants
  2-year survival: Alive | 25
  2-year survival: Deceased | 3
  5-year survival: Alive | 20
  5-year survival: Deceased | 8
  10-year survival: Alive | 12
  10-year survival: Deceased | 16
  Overall survival: Alive | 7
  Overall survival: Deceased | 21

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was collected and assessed every 6 months via phone and then via medial record review during long-term follow-up, up to 14 years, AEs collected and recorded at least 4 weeks (30 days) after the last exposure to the study drug (up to day 90).
Arm/Group | Adenovirus/PSA Vaccine
All-Cause Mortality (participants affected / at risk) | 21/32
Serious Adverse Events (participants affected / at risk) | 3/32
Other Adverse Events (participants affected / at risk) | 18/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adenovirus/PSA Vaccine (N=32)
Pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstruction/stenosis of airway - Bronchus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adenovirus/PSA Vaccine (N=32)
Headache (General disorders) | 4 (4)
Injection site irritation (Skin and subcutaneous tissue disorders) | 4 (4)
Cold and flu symptoms (General disorders) | 5 (5)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-01-27): https://cdn.clinicaltrials.gov/large-docs/24/NCT00583024/Prot_SAP_000.pdf
  • Informed Consent Form (2013-04-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT00583024/ICF_001.pdf